CLINICAL TRIAL: NCT00695123
Title: Screening of Subjects to Determine Eligibility to Safely Participate in Blood Disorders Studies
Brief Title: Screening for Subjects to Participate in Studies of Blood Disorders
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080156; 08-H-0156
Record Dates: First submitted 2008-06-07; First posted 2008-06-11 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Bone Marrow Transplant; Sickle Cell Disease; G-CSF
Keywords: Bone Marrow Transplant; Sickle Cell Disease; G-CSF; Apheresis
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Only 1 participant group (cohort): The subject may have a blood disorder, may be a stem cell transplant donor, or may be a healthy volunteer.

SUMMARY:
This study will determine eligibility for participation in research studies on blood disorders conducted by the National Heart, Lung and Blood Institute and the National Institute of Diabetes, Digestive, and Kidney Diseases.

Healthy volunteers, patients with blood disorders under study by NHLBI and NIDDK and potential stem cell donors for patients with blood disorders who are 8 years of age and older may be eligible for this screening protocol. (Healthy volunteers who qualify for research protocols would serve as control subjects.)

Participants undergo the following tests and procedures:

Healthy Volunteers

* Medical history, physical examination, blood tests and urine sample collection.
* Buccal mucosa sample collection. (Cells are collected from the inside of the cheek by gentle scraping with a bristly brush.)
* Bone marrow aspiration (only for volunteers 18 years of age and older).

Potential Stem Cell Donor

-Same as for healthy volunteers plus evaluations that may include electrocardiogram, echocardiogram, imaging studies (X-rays, CT scans, MRI scans and others), heart evaluation, and lung function tests.

Patient with Blood Disorder

* Same as for stem cell donors plus additional evaluations and treatments that may include radiation oncology evaluation, catheter placement, blood transfusions, kidney and liver biopsies. Short courses of drug treatment for induction of fetal hemoglobin in sickle cell patients, and/or iron chelation in patients receiving chronic red cell transfusions may be included as well.

DETAILED DESCRIPTION:
This study allows the evaluation of subjects in order to determine their ability to safely participate in other active NIH research studies studying blood disorders. This protocol serves several purposes: 1) allows detailed investigations into the blood disorders of these subjects, and the status of other organ systems that would determine their ability to safely tolerate specific aspects of active research protocols; 2) allows investigators to offer clinical diagnostic testing and procedures to patients if this treatment will facilitate their participation in a clinical trial; 3) allows investigations as to whether a donor is HLA matched, fit to receive G-CSF, and fit to undergo apheresis and therefore eligible to participate as a donor on a bone marrow transplant protocol; 4) allows the evaluations of healthy volunteers as to whether they are eligible for participation as control subjects on protocols that require generally good health status by history or physical exam findings, or laboratory assessments; and 5) allows for the collection and storage of research specimens and samples obtainable by minimal risk for development or validation of novel clinical tools and approaches to disease. After completion of the screening process, the subject will either be offered a chance to participate in an active research protocol, or if no appropriate protocol is identified, subjects with blood disorders will have recommendations for other treatment options relayed to them and/or to the primary or referring physician.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be entered on this protocol at the time of their first visit to the NIH Clinical Center outpatient clinic or inpatient service if the subject is able to give consent/assent and the subject may have a blood disorder, may be a stem cell transplant donor, or may be a healthy volunteer.

* The subject or the subject s guardian is capable of informed consent and willing to sign the consent form after initial counseling by clinical staff. Additional consent for clinically indicated procedures (central venous catheter placement; biopsy of liver, kidney; or bone marrow) or blood transfusions will be obtained.
* The subject has a reasonable likelihood of having a disorder for which MMB or MCHB has an active research protocol, and based on information received from an outside physician, he/she appears to meet at least preliminary eligibility criteria for that protocol.
* The subject has been identified as a potential donor for a subject for whom the MMB or MCHB has an active stem cell transplant protocol and based on information received from an outside physician, he/she appears to meet preliminary eligibility as a donor.
* The subject (age greater than or equal to18) is a healthy volunteer for whom the MMB or MCHB has an active study recruiting healthy normal volunteers and he/she appears to meet preliminary eligibility as a healthy volunteer.

EXCLUSION CRITERIA:

* Unable to comprehend the investigational nature of the protocol participation
* Abnormal CBC for healthy volunteers
* Positive pregnancy test for stem cell donors and healthy volunteers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be entered on this protocol at the time of their first visit to the NIH Clinical Center outpatient clinic or inpatient service if the subject is able to give consent/assent, and the subject may have a blood disorder, may be a stem cell transplant donor, or may be a healthy volunteer.
Sampling Method: Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2008-07-03 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Evaluate consented subjects with blood disorders | ongoing
  1) to assess the hematologic problems, the status of other organ systems, and their ability to safely tolerate active treatment protocols; 2) to determine eligibility for active MMB and/or MCHB protocols. Subjects may require screening procedures and clinical treatments in order to determine eligibility for participation; and 3) to allow time for counseling and deliberation regarding best treatment option

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Hsieh, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2008-H-0156.html